CLINICAL TRIAL: NCT03839017
Title: Impact on Performance of the Use of a Digital Cognitive Aid in Simulated Crisis and Stress Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEJKA Jean-Christophe (Other)
Responsible Party: Sponsor-Investigator, CEJKA Jean-Christophe, Teaching Hospital Practitioner, Claude Bernard University
Organization: Claude Bernard University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIMMAXMARCHERYAN2
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: War Injury
Keywords: Forward medicalization; Cognitive aid; Crisis situation; High-fidelity simulation; Performance

STUDY DESIGN:
Intervention Model Description: With or without the cognitive aid
Who Masked: Participant
Masking Description: Single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive aid (Experimental): The leader uses a digital cognitive aid designed as a smartphone app during advanced combat casualty care. Intervention: Device: SIMMAXMARCHERYAN2 Digital cognitive aid during the management of simulated war wounded.
  Interventions: Device: SIMMAXMARCHERYAN2
- Without digital cognitive aid (Experimental): The leader practices advanced combat casualty care without the digital cognitive aid designed as a smartphone app. Intervention: Device: SIMMAXMARCHERYAN2 Without digital cognitive aid during the management of simulated war wounded.
  Interventions: Device: SIMMAXMARCHERYAN2

INTERVENTIONS:
Device: SIMMAXMARCHERYAN2 — Digital cognitive aid during the management of simulated war wounded.

SUMMARY:
The previous investigators' studies (MAX, Lelaidier et al, BJA 2017, & SIMMAXMARCHERYAN) clearly showed that the use of a digital cognitive aid in the hand of the leader significantly improves the management of anaesthesia and intensive care emergencies as well as basic combat casualty care.

The present study exclusively deals with the advanced management of simulated combat casualties by military doctors and nurses using the same digital cognitive aid adapted for MARCHE RYAN algorithm.

DETAILED DESCRIPTION:
The epidemiology of battlefield mortality highlights the need for safety and speed of care in an environment under very high stress. Indeed, it has been found that about 90% of those killed in action die before reaching the first hospital or care unit. Management algorithms such as ABCDE, SAFE MARCHE RYAN and local protocols are among the many doctrines to be applied by military health professionals when dealing with serious trauma in emergencies in different practice settings. During combat, their actions are carried out under enemy fire, in darkness, in extreme environments, for a significant number of victims and with limited means. As a result, on the battlefield, this multitude of choices and specific conditions of practice can make it difficult to apply the guidelines for the management of war-wounded in critical and stressful situations and can be a source of medical error. Health simulation is one of the main tools for training and preparation in a safe environment for unsafe situations ("never the first time on the patient"). A new decision-making and protocolization tool is available for health professionals: the MAX (Medical Assistant eXpert) cognitive aid, which has already proven its effectiveness in reducing the number of errors in the management of vital distress in anesthesia and in basic combat casualty care.

Materials and Methods:

Population studied: military doctors and nurses from the forces, both male and female, of varying ages and operational experience, planned to be deployed on External Operations (OPEX) or Short-term Mission (MCD), designated by the Val-de-Grâce School as learners for the " Survival Conditioning of the War Wounded " (MCSBG) continuing training course.

Study design (conduct): analytical, prospective, randomized, controlled, unblinded study conducted during the MCSBG training courses as part of the operational preparation of military doctors and nurses of the forces within the Center for Education and Simulation in Operational Medicine (CESimMO) in Toulon. The investigators had four pairs of learners work on one afternoon during each week-long training session. Each pair of learners completed two different scenarios of similar difficulty and complexity. Four blocks of scenarios were defined on which the pairs were able to work. The pairs were initially randomly assigned to two groups: Group 1 where the first scenario was performed with the MAX CA and Group 2 where the CA was used in the second scenario. Each group therefore performed a simulated scenario with and without MAX. The scenarios used either high-fidelity mannequins (SimMan 3G / ALS, Laerdal, Stavanger, Stavanger, Norway) or hybrid standardized patients (standardized subjects equipped with anatomical prostheses that allowed their management including technical procedures).

MAX CA Description: MAX is a digital AC, developed by J.C. CEJKA, and initially intended for the management of anesthesia and resuscitation emergencies. For the MARCHE RYAN protocol, each action was presented sequentially by the CA and had to be validated before the next one was displayed (READ and DO mode). It was possible to go back in order to review the validated actions and at the end of the procedure, the user had the possibility to make a final check of all his actions. The evaluation of the effectiveness of MAX was previously carried out at the Lyon center for teaching through health simulation (CLESS, UCBL1 - Claude Bernard University Lyon 1), but also during the training of Medicalization in hostile environments (MEDICHOS) and the continuing training in 2nd level combat rescue / casualty care (SC).

Use of the AC MAX in the study: Each participant disposed of a MAX application when dealing with war wounded in simulated situations. The presentation of the application and its handling was done on the first morning of each course, and a license for downloading and using the application was granted to each participant. The instructors were present to answer any questions about this CA. The anonymity of the study participants was ensured and their volunteering as well as the authorization to take pictures and use the videos collected at the beginning of each course.

Participants were requested to absolutely use the application for one of the two scenarios (randomized choice). The fact of being able to use MAX was communicated to them each time during the scenario briefing. More precisely, the one running the MARCHE RYAN algorithm had to use the MAX AC for a complete sequence, from the beginning of the scenario and follow MAX's prompts until the end of the protocol. The participants decided who in the pair will use MAX, however this person had to use both MAX+ and MAX- scenarios according to the MARCHE RYAN protocol. One of the instructors/facilitators who followed this process was to remind them of this requirement during the care of war wounded when necessary, and to impose the use of CA, if applicable.

Randomization by block allocation was performed using open source software R (randomizr library, R Foundation for Statistical Computing, Vienna, Austria, version 3.4.1), to have a homogeneous distribution of participants in Group 1 (MAX first) and Group 2 (MAX second), according to four blocks (1 block per scenario passage). The types of scenarios, the locations where the training took place and the distribution of trainers were the same for all MCSBG courses included in the study. The designation of the pairs was made on the first day of each course by the trainers in title of the CESimMO of Toulon, from the list of trainees participating.

The calculation of the number of subjects required was carried out a priori on the basis of data from the work of R. Lelaidier and M. Truchot studying the effect of MAX CA on technical and non-technical performance. In this work, the scenarios being of similar difficulty, investigators do not expect any significant effect from this factor, so the differences in means will be influenced by the use of MAX. The size of the expected effect was calculated from a mean difference of 13 points, and a standard deviation of sd=11, with n=8 groups (4 scenario blocks with or without MAX), which equates to a MAX CA effect size of 0.4 between the eight groups. The recruitment of 32 pairs will allow investigators to have a power of 0.88 with a first species risk of 0.05. In other words, a population of 32 pairs will allow investigators to show a minimum effect size of f=0.35, with a power of 0.8 and a first species risk of 0.05. There was no interim analysis planned for this study.

Data collection and analysis:

All performances were filmed (using GoPro Hero 4 cameras, San Mateo, California, USA) and anonymized. Each video recording of the MAX+ and MAX- scenarios was remotely rated by two independent evaluators (NP and PR), using the technical and non-technical performance rating grids. The scales used have already been published in international journals. If a difference of more than one point out of 10 was found between the two ratings, a third assessor (AP) would act as mediator.

A questionnaire (quiz) was also distributed to participants at the end of each course to find out how they felt about the influence of the use of the AC MAX on their performance.

ELIGIBILITY:
Inclusion Criteria:

* Military doctors and Nurses
* Under initial or continuous training of Combat Casualty Care 3rd level
* Agreed to use the cognitive aid

Exclusion Criteria:

* Doesn't agree to use the cognitive aid

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Technical Performance: percentage of actions and steps in the MARCHE RYAN protocol performed by each subject with or without the CA MAX | Time 0-30 minutes
  As compared to a Reference Task List including between 11 and 16 critical actions to be performed. This grid was used to rate technical performance in each scenario. Each action was recorded: 0 (action not performed), 1 (action performed at the wrong time, with the wrong dosage or inaccurately) or 2 (action performed correctly and at the right time). The individual scores were summed and transformed into a percentage of the maximum achievable score.
  Statistical analysis and calculation of the number of pairs required:
  The analysis of the effect of the use of MAX CA on learners' technical performance will be carried out using a 3-factor repeated-measure ANOVA: the use of MAX, the scenario, and whether the scenario is played first or second. A post-hoc analysis by the Bonferroni test will be carried out to compare the groups.

SECONDARY OUTCOMES:
Non technical skills performance measured using the TEAM scale, MAX+ vs MAX- | Time 0-30 minutes
  As measured by the TEAM scale score. Each of the 11 skills was rated between 0 and 4, and the overall performance between 1 and 10, for a maximum total of 54 points. Non-technical performance could therefore vary between 1 and 54.

CONTACTS AND LOCATIONS:
Overall Officials: Jean J Lehot, MD, PhD, Study Director — Claude Bernard University
Locations (1):
- CESimMO, Toulon, PACA, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paraschiv AP, Cejka JC, Lilot M, Aigle L, Lehot JJ, Balanca B. Impact of a Digital Cognitive Aid on the Performance of Military Healthcare Teams During Critical Care Management in a Warfront Injury Situation: A Simulation Randomized Controlled Study. Simul Healthc. 2022 Jun 1;17(3):163-169. doi: 10.1097/SIH.0000000000000623. Epub 2021 Dec 15. PMID 34934026
- See also: Précloux P, Wey P-F, Bérend M. et al. Opération " Pamir " : bilan et analyse de l'activité des postes médicaux de Rôle 1 à partir du Registre santé de l'avant pour l'année 2011. Médecine et Armées 2014, 42, 4: 299-308 — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=2ahUKEwj78-W3k7HgAhVQcZoKHV3BB_oQFjAAegQIARAC&url=http%3A%2F%2Fwww.ecole-valdegrace.sante.defense.gouv.fr%2Fcontent%2Fdownload%2F5262%2F66195%2Ffile%2F02%2520Precloux%2520P.%2520Operation%2520Pamir%2520bilan%2520et%2520analyse%2520activite%2520des%2520postes%2520medicaux%2520role%25201%2520RSA%25202011.%2520Medecine%2520et%2520Armees%25202014-4.%2520299-309..pdf&usg=AOvVaw3yJGF-F9y6y0NrjPdLdnN_
- See also: Hoffmann et al. Épidémiologie des blessés de guerre français en Afghanistan : de la blessure à la réinsertion. Urgences 2015 - Congrès de la Société Française de Médecine d'Urgence, At Paris, Volume : Chapitre 83 — https://www.researchgate.net/publication/279559442_Epidemiologie_des_blesses_de_guerre_francais_en_Afghanistan_de_la_blessure_a_la_reinsertion
- See also: Holcomb JB. Major scientific lessons learned in the trauma field over the last two decades. PLoS Med 2017, 14(7): e1002339 — https://doi.org/10.1371/journal.pmed.1002339
- See also: Holcomb JB, Stansbury LG, Champion HR et al. Understanding casualty care statistics. 2006, Repéré à PubMed.gov. DOI : 10.1097/01.ta.0000203581.75241.f1 — https://europepmc.org/abstract/med/16508502
- See also: Jones C, Bond C. 68W. Advanced Field Craft. Combat Medic Skills. 2010, AAOS (American Academy of Orthopaedic Surgeons). Jones and Bartlett Publishers USA — https://books.google.fr/books?id=7eoDZyAL3XcC&pg=PR4&lpg=PR4&dq=Jones+C,+Bond+C.+68W.+Advanced+Field+Craft.+Combat+Medic+Skills.+2010,+AAOS+(American+Academy+of+Orthopaedic+Surgeons).+Jones+and+Bartlett+Publishers+USA&source=bl&ots=vVeVUklZRO&sig=ACfU3U2-dgXhA3CsuumrYA3a0mAoALHkpA&hl=fr&sa=X&ved=2ahUKEwj1nfG4lbHgAhXb8qYKHR-BCJEQ6AEwAXoECAkQAQ#v=onepage&q=Jones%20C%2C%20Bond%20C.%2068W.%20Advanced%20Field%20Craft.%20Combat%20Medic%20Skills.%202010%2C%20AAOS%20(American%20Academy%20of%20Orthopaedic%20Surgeons).%20Jones%20and%20Bartlett%20Publishers%20USA&f=false
- See also: École du Val-de-Grâce. Enseignement du Sauvetage au Combat. 2012 — https://sofia.medicalistes.fr/spip/IMG/pdf/Enseignement_du_Sauvetage_au_Combat-_Referentiel_de_formation_janvier_2012_.pdf
- See also: McSwayn NE, Butler FK. Prehospital Trauma Life Support. Military Seventh Edition. 2011, Mosby Jems Elsevier USA — https://www.elsevier-masson.fr/?gclid=Cj0KCQiAtP_iBRDGARIsAEWJA8iexeQLMqpyg_F5nJoPgI8ykzsLofLrC6MZNG0fGWNX1L07r3fmJIgaApPPEALw_wcB
- See also: Selye H. Le stress de la vie. Le problème de l'adaptation 1975. Gallimard, coll. " L'avenir de la science ", 2e édition — http://www.gallimard.fr/Catalogue/GALLIMARD/Les-Essais/Le-Stress-de-la-vie
- See also: Morgenstern J. Performance Under Pressure. Psychology 2017, 24 (2) : 168-88 — https://www.ncbi.nlm.nih.gov/pubmed/27981877
- See also: Boet S, Granry J-C, Savoldelli G. La simulation en santé. De la théorie à la pratique. 2013, Springer-Verlag France — https://link.springer.com/book/10.1007/978-2-8178-0469-9
- See also: Lelaidier R, Balança B, Boet S, Faure A, Lilot M, Lecomte F, Lehot J-J, Rimmelé T, Cejka J-C. Use of a hand-held digital cognitive aid in simulated crises: the MAX randomized controlled trial. BJA, Nov. 2017, vol. 119, 5 : 1015- — https://www.ncbi.nlm.nih.gov/pubmed/29028930
- See also: Marshall S D. Lost in translation? Comparing the effectiveness of electronic-based and paper-based cognitive aids. British Journal of Anaesthesia, Oct. 2017, 0 (0): 1-3 — https://www.ncbi.nlm.nih.gov/pubmed/29028936
- See also: Lehot J J, Le Goff A, Wegrzyn J, Barthelemy-Bougault J, Wey P-F, Cavallo J-D. Enseignement par simulation : un exemple de coopération civilo-militaire. Médecine et Armées 2017, 45, 5 : 611-616 — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=2ahUKEwiI9JSAl7HgAhVIxKYKHaT2B0sQFjAAegQIBhAC&url=http%3A%2F%2Fwww.ecole-valdegrace.sante.defense.gouv.fr%2Fcontent%2Fdownload%2F7825%2F84385%2Ffile%2F14%2520Lehot%2520JJ.%2520Enseignement%2520par%2520simulation.%2520Exemple%2520de%2520coop%25C3%25A9ration%2520civilo-militaire.%2520M%25C3%25A9decine%2520et%2520Arm%25C3%25A9es%2520s%25202017-5-611-6.pdf&usg=AOvVaw1rpcYQWWJ-0UVdGy7tH8pl
- See also: Cooper S, Wakelam A. Leadership of resuscitation teams: 'Lighthouse Leadership'. Resuscitation 1999; 42: 27-45 — https://www.ncbi.nlm.nih.gov/pubmed/10524729
- See also: Cooper S, Cant R, Connell C, Porter J E, Symmons M, Nestel D, Liaw S Y. Measuring teamwork performance: Validity testing of the Team Emergency Assessment Measure (TEAM) with clinical resuscitation teams. Resuscitation 2016; 101: 97-101 — https://www.ncbi.nlm.nih.gov/pubmed/26875992